CLINICAL TRIAL: NCT06989879
Title: Knowledge of Students About Vitamin A and Assessment of Eye Manifestations in Quranic Schools (Khalwai) Khartoum State, Sudan 2022
Status: Completed | Type: Observational
Sponsor: University of Khartoum (Other)
Responsible Party: Principal Investigator, Elkhidir Bashir Elkhidir Ali, Principal investigator, University of Khartoum
Other Study IDs: COMMED 2022-94-14
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Vitamin A Deficiency; Night Blindness
Keywords: Vitamin A deficiency; Night blindness; Quranic boarding school; knowledge; nutrition
MeSH Terms: conditions — Vitamin A Deficiency; Night Blindness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study that aims to study vitamin A deficiency status, knowledge, and nutritional assessment among Khalwa (Quran boarding school) individuals. we want to assess the magnitude of the problem and put appropriate recommendations for it.

ELIGIBILITY:
Inclusion Criteria:

* All Khalwa (Quranic-boarding-school) dormitory residents of in East-Nile province, Khartoum State

Exclusion Criteria:

* Anyone who refuses to participate in the study.
* Those who live with their families

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Khalwa (Quranic boarding school) dormitory residents are either dedicated teachers, students, or those who teach and study at the same time. The study participants were those who lived in the dormitory regardless of their status. Those in the last category were counted as students.
  The study was conducted in traditional Quran centers in East Nile Province, Khartoum.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence rate of night blindness | At enrollment
Vitamin A knowledge score | At enrollment
Prevalence rate of vitamin A deficiency signs | At enrollment
Prevalence rate of respiratory tract infection | At enrollment
Prevalence rate of diarrhea | At enrollment
Food specific (milk, vegetables, fruits, etc.) prevalence rate of eating/drinking from outside dormitory | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Khartoum, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes